CLINICAL TRIAL: NCT04439669
Title: Complex Regional Pain Syndrome - Diagnostics, Pathophysiological Mechanisms, and Response to Treatment With Noninvasive Brain Stimulation
Brief Title: CRPS - Diagnostics, Pathophysiological Mechanisms, and Response to Treatment With Noninvasive Brain Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Hanna Harno, Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TYH20162222
Record Dates: First submitted 2020-03-31; First posted 2020-06-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Transcranial Magnetic Stimulation; Complex Regional Pain Syndrome of Upper Limb (Disorder)
Keywords: TMS; CRPS; pain; fMRI; quality of life; mood; cognitive function; DNA
MeSH Terms: conditions — Reflex Sympathetic Dystrophy; Pain

STUDY DESIGN:
Intervention Model Description: The patients are first randomized to receive either sham stimulation or right "S2" for three week period (10 stimulation sessions). Thereafter, a 3 month followup period (clinical checkup at a research visit at 1 month, RN structured telephone interviews at 2 and 3 months). If pain ≥5/10 at 3 month interview, the patient is offered an open label nrTMS treatment phase, in which the protocol depends on the first protocol of the RCT phase.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant does not know whether the stimulation is sham or active. The doctor or nurse giving the stimulation knows the target and whether the stimulation is sham or active. The RN and the clinician (conducting screening and 1 month clinical visit) do not know the stimulation type or target until month 3, when the code is opened.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Starts with active stimulation (Active Comparator): Active nrTMS is given to "S2" at the right side (10 sessions in a three week period). Thereafter, a new, open label phase will start if the average pain at 3 month follow-up is ≥5/10. Then, the nrTMS will be targeted to M1 contralateral to the side of pain. After 5 stimulation sessions the response is evaluated. If pain is still ≥510, the investigators change the target to the "S2" on the left side for five sessions. If there is response with pain relief, a maintenance therapy with this target is offered for 6 months with gradually reducing stimulation sessions.
  Interventions: Device: Active nrTMS and open phase
- Starts with sham stimulation (Placebo Comparator): Sham nrTMS will be targeted to the "S2" on the right side, but using a sham box/coil. Stimulation period is similar than for the active comparator. Similarly, thereafter, a new, open label phase will start if the average pain at 3 month follow-up is ≥5/10. Then, the nrTMS will be targeted to "S2" at the right side. After 5 stimulation sessions the response is evaluated. If pain is still ≥5/10, the investigators change the target to M1 on the contralateral side of the pain and furthermore to "S2" at the left side after 5 stimulation sessions, if pain is still ≥5/10.
  Interventions: Device: Sham nrTMS and open phase

INTERVENTIONS:
Device: Sham nrTMS and open phase — Navigated repetitive TMS treatment (10 sessions during a three-week period) randomized to sham. In the following open phase stimulation the treatment targets are the right "S2"-contralateral M1-left "S2".
  Other Names: Starts with sham stimulation
  Arms: Starts with sham stimulation
Device: Active nrTMS and open phase — Navigated repetitive TMS treatment (10 sessions during a three-week period) randomized to "S2". In the following open phase stimulation the treatment targets are contralateral M1 and left "S2". If the patient benefited from active "S2" stimulation, but the treatment effect faded in follow-up, the open phase stimulation starts with right "S2".
  Other Names: Starts with active stimulation
  Arms: Starts with active stimulation

SUMMARY:
This is a sham controlled, randomized, double-blind, navigated repetitive Transcranial Magnetic Stimulation (nrTMS) study for the treatment of complex regional pain syndrome (CRPS types 1 and 2). The investigators study factors that may contribute to development, maintenance, or treatment responses with clinical, sleep, and psychiatric questionnaires and clinical examinations, quantitative sensory testing and neurophysiologic recordings, genetics, and MRI techniques.

DETAILED DESCRIPTION:
rTMS hypothetically disrupts the default networks related to chronic pain and renders the brain more susceptible to drugs, rehabilitation, or cognitive behavioral therapy. In addition, there is experimental evidence that rTMS releases factors that are involved in endogenous top-down modulation of pain and neural plasticity. Thus, the analgesic effect of rTMS may be mediated via enforcing endogenous pain control systems at the brain level, in addition to its effects on neuroplastic effects.

For active, navigated stimulation targets the investigators have the parietal opercular cortex overlying the secondary somatosensory cortex ("S2") and the primary motor cortex (M1).

The investigators randomize participants to first receive nrTMS to the right "S2" or sham stimulation. After ten sessions the investigators follow up the participants up to three months. At three months, if the average pain is ≥5/10 in numeric rating scale (NRS), the participant is offered an active, open nrTMS treatment phase depending on which treatment the participant first received. If the participant benefits from the open label treatment, a maintenance therapy is offered (6 months with gradually reducing nrTMS treatment frequency). The symptoms and quality of life are followed with questionnaires and diaries. After the maintenance period, the RN calls a structured interview at 1, 3, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* CRPS 1 or 2 of the upper limb
* Duration ≥ 6 months
* Mean pain (NRS) intensity ≥5/10
* Medical and other therapies have failed

Exclusion Criteria:

* Other stimulation therapies apart from transcutaneous nerve stimulation
* psychotic disorder
* severe depression
* use of strong opioids
* epilepsy
* any contraindication for MRI
* abuse of alcohol or drugs
* ongoing insurance or other entitlement cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-08-28 (Actual); Primary Completion 2021-07-29 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
15-item quality of life measure | Change from baseline at one month
  Quality of life (15D questionnaire) with 15 question items with 5 alternatives in each. The scores range between 15 to 75 with 15 the best and 75 the worst quality of life.

SECONDARY OUTCOMES:
Mean pain intensity and interference | Baseline, during stimulation, and two weeks after the intervention
  Numeric rating scale (NRS, 0= no pain and 10= the worst pain imaginable)
Weekly pain intensity and interference | Up to 3 months after intervention
  Pain questionnaires (numeric rating scale (NRS, 0= no pain and 10= the worst pain imaginable)
Sleep interference and quality | Baseline and 1,2,and 3 months after intervention
  Insonnia severity index (ISI). There are seven questions with scale 0 to 4 (0 with no symptoms and 4 with the worst symptoms). The scores are added up to get a total score ranging from 0 to 28. A higher score means a worse outcome.
Clinical neurophysiology measures | Baseline and one week after intervention
  Quantitative sensory testing (QST) with standardized reporting
Cognitive assessment A | Baseline and one month after the intervention
  Cognitive function assessment by Cogstate, a computer based detection and identification task. Answers yes or no, standard reporting.
Hand strength | Baseline and one week after the intervention.
  Hand motor function measured e.g. by Jamar (kg)
Biochemical tests | At baseline
  Blood samples: inflammatory markers (e.g. high sensitivity CRP, proteomics). Standard reporting
Brain imaging: Default mode networks | Baseline and one week after intervention
  Resting state fMRI
CRPS symptom severity | Baseline and at one month
  CRPS severity scale (CSS, 0=no symptoms or signs, 17=maximum score with symptoms and signs)
Patient global impression of change | 1, 2, and 3 months and through study completion, an average of 1 year
  Global impression of change (GIC, 1=very much improved, 7= very much worse)
Screening of psychiatric symptoms and diagnostics | Up to 24 weeks
  Psychiatric interveiw (SCID II) with symptom and diagnostic description. Nine questions, answers yes or no, standard reporting. The more "yes"-answers, the worse the outcome.
Hand mobility | Baseline and one week after intervention
  Angles of the joints in the hand (degrees)
Cognitive assessment B | Baseline and one month after the intervention
  Wechsler Memory Scale III (WMS-III) subtest: digit span. Number of digits recalled. Standard reporting.
Cognitive assessment C | Baseline and one month after the intervention
  Wechsler Memory Scale III (WMS-III) subtest: word list. Number of words recalled. Standard reporting.
Cognitive assessment D | Baseline and one month after the intervention
  Bourdon-Wiersma (Attention and concentration): number of visual stimuli found.
Cognitive assesment E | Baseline and one month after the intervention
  Trail-Making Test (Parts A and B): time spent (seconds) for visual scanning task. Standard reporting.
DNA | At baseline
  DNA analysis. Standard reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Eija Kalso, Professor, Study Chair — Helsinki University Hospital, Pain Clinic; Satu Jääskeläinen, Professor, Study Chair — Turku University Hospital, Dept. of Clinical Neurophysiology; Hanna Harno, MD, PhD, Study Director — Helsinki University Hospital, Pain Clinic
Locations (2):
- Finland (2):
  - Turku University Hospital, Pain Clinic, Turku, Southwest Finland
  - Helsinki University Hospital, Pain Clinic, Helsinki, Uusimaa

IPD SHARING:
Plan to Share IPD: No
The Ethics committee doesn't allow that due to privacy agreements.

REFERENCES:
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Jaaskelainen SK, Lindholm P, Valmunen T, Pesonen U, Taiminen T, Virtanen A, Lamusuo S, Forssell H, Hagelberg N, Hietala J, Pertovaara A. Variation in the dopamine D2 receptor gene plays a key role in human pain and its modulation by transcranial magnetic stimulation. Pain. 2014 Oct;155(10):2180-7. doi: 10.1016/j.pain.2014.08.029. Epub 2014 Aug 29. PMID 25180011
- [Derived] Liesto S, Aho T, Jaaskelainen SK, Hietanen M, Kalso E. Cognitive Function in Patients With Complex Regional Pain Syndrome (CRPS). Eur J Pain. 2025 Jul;29(6):e70070. doi: 10.1002/ejp.70070. PMID 40626344